CLINICAL TRIAL: NCT06497413
Title: Brain Vascular and Neurocognitive Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Matthew Brothers, Professor, The University of Texas at Arlington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-0011
Record Dates: First submitted 2024-06-10; First posted 2024-07-11 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Decline; Cognitive Dysfunction; Alzheimer Disease; Vascular Disease, Peripheral
Keywords: cerebral oxygenation; cognitive function; brain blood flow
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Individuals will be randomly assigned either an experimental or a control condition
Who Masked: Investigator
Masking Description: The investigators will use a randomizer to assign the participant with either the experimental or sham treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcranial Photobiomodulation (Experimental): Transcranial Photobiomodulation (tPBM) is a novel and non-invasive strategy that utilizes a helmet that delivers low-level laser therapy to activate intracellular enzymatic pathways leading to an increase in mitochondrial activity, cerebral oxygenation, and thus neural and overall brain function. Importantly, this approach improves cognitive function in various animal models and limited human populations. Furthermore, there is limited evidence to suggest that these neurocognitive improvements are in-part related to increases in cerebral blood flow and cerebral vascular function/health.
  Interventions: Device: Transcranial Photobiomodulation
- Sham condition (Placebo Comparator): In this condition the participants will wear the Transcranial Photobiomodulation (tPBM) headgear; however, no light will be delivered.
  Interventions: Device: Transcranial Photobiomodulation helmet (Neuradiant 1070 Plus) with no light administered

INTERVENTIONS:
Device: Transcranial Photobiomodulation — The transcranial photobiomodulation will be delivered through the Neuradiant 1070 Plus-Programmable 4-Quadrant Photobiomodulation System. This is a commercially available helmet that will be purchased from a commercially available source.
  Arms: Transcranial Photobiomodulation
Device: Transcranial Photobiomodulation helmet (Neuradiant 1070 Plus) with no light administered — In this condition the participants will wear the Transcranial Photobiomodulation helmet (Neuradiant 1070 Plus); however, the light will not be administered.
  Arms: Sham condition

SUMMARY:
The overall research objective of this proposal is to determine the acute and chronic impact of transcranial photobiomodulation on indices of cerebral vascular health and neurocognitive function.

DETAILED DESCRIPTION:
Neurocognitive conditions and diseases including cognitive dysfunction, Alzheimer's disease and related dementias (ADRD) are among the fastest growing causes of morbidity and mortality. ADRDs impact > 5 million people in the United States alone and > 47 million people worldwide. The physiological reasons for these conditions are multifactorial but one contributing factor is impaired cerebral vascular function/health. Importantly, impaired cerebral vascular function/health results in cerebral hypoperfusion thereby contributing to neuronal damage and neurodegenerative processes ultimately contributing to the aforementioned neurocognitive impairments. Furthermore, it is critical to investigate therapeutic strategies to combat this elevated risk. One promising approach is Transcranial Photobiomodulation (tPBM) which is a novel and non-invasive strategy that utilizes low-level laser therapy to activate intracellular enzymatic pathways leading to an increase in mitochondrial activity, cerebral oxygenation, and thus neural and overall brain function. Importantly, this approach improves cognitive function in various animal models and limited human populations. Furthermore, there is limited evidence to suggest that these neurocognitive improvements are in-part related to increases in cerebral blood flow and cerebral vascular function/health. However, information regarding the mechanisms and effectiveness of tPBM are still relatively unknown - which represents a critical knowledge gap in the literature.

Therefore, the overall research objective is of this proposal is to determine the impact of tPBM on indices of neurocognitive and cerebral vascular health. The following objectives / aims will be explored:

1. Primary Aim - The primary endpoint is the effect of acute (i.e. one-time) and repeated (i.e. up to 8 times in a 4-week period) exposure to tPBM on outcomes associated with elevated risk for various neurocognitive and pathophysiological conditions/diseases. These outcomes include neurocognitive function and indices cerebral blood vessel function/health.
2. It is hypothesized that both acute and repeated exposure to tPBM will have a beneficial impact on the outcome variables of neurocognitive function and indices cerebral blood vessel function/health.

ELIGIBILITY:
Inclusion Criteria:

* Both men and women between the ages of 18-80 and of any race/ethnicity will be included in this study.

Exclusion Criteria:

* Individuals who have donated more than 550 ml of blood within the past 8 weeks will not have blood drawn from them in this protocol. However, if they remain interested in the study, and otherwise meet the inclusion criteria, then the investigators may still opt to proceed with data collection.
* Abnormal results from the blood screening will not impact eligibility for the study.
* Individuals with brain injuries/surgeries in a year before the study and individuals who can not provide consent on their own will be excluded from participation.
* Pregnant subjects, women who are breast feeding, and children (i.e. younger than 18) will not be recruited for the study. This will be assessed via self-report.
* If a subject has any allergies to spandex/lycra, the subject will be excluded. However, latex allergies are not contraindicated.
* Individuals with cardiac pacemakers and/or implantable cardioverter defibrillators and individuals with epilepsy will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
Cerebral vasodilator function | Immediately before the start of the experimental or sham condition intervention. And immediately after the end of the experimental or sham condition intervention.
  This will be assessed as the increase in blood flow in the middle cerebral artery during a hypercapnic stimulus
Neurocognitive function | Immediately before the start of the experimental or sham condition intervention. And immediately after the end of the experimental or sham condition intervention.
  This will be assessed using the NIH Toolbox which is a battery that consists of several cognitive challenges.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Brothers, PhD, Principal Investigator — University of Texas at Arlington
Locations (1):
- UT Arlington - Science and Engineering Innovation and Research Building, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No There is not a plan to share individual participant data (IPD)